CLINICAL TRIAL: NCT07083635
Title: Transdermal Ethinyl Estradiol and Norelgestromin for Treating Irregular Vaginal Bleeding in Contraceptive Implant Users: A Randomized, Double-Blind, Controlled Trial
Brief Title: Transdermal Ethinyl Estradiol and Norelgestromin for Irregular Bleeding in Contraceptive Implant Users
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Tunchanok Juntamongkol, MD, Principal Investigator, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 107/68
Record Dates: First submitted 2025-07-13; First posted 2025-07-24 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Menstruation Disturbances; Metrorrhagia; Uterine Hemorrhage; Contraception Behavior
Keywords: Contraceptive implant; Abnormal vaginal bleeding; Bothersome vaginal bleeding; Irregular vaginal bleeding; Transdermal hormonal contraception; Ethinyl estradiol; Norelgestromin; Abnormal uterine bleeding; Contraceptive-induced bleeding; Combined hormonal contraception; Hormonal contraceptive patch
MeSH Terms: conditions — Menstruation Disturbances; Metrorrhagia; Uterine Hemorrhage; Contraception Behavior | interventions — Ethinyl Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Transdermal Hormonal Contraceptive Patch (Ethinyl Estradiol and Norelgestromin)
  Active Ingredients:
  Ethinyl Estradiol: 600 micrograms per patch Norelgestromin: 6 milligrams per patch
  Administration Schedule:
  1 patch applied every 7 days Total treatment duration: 21 days (3 patches total) Application Site: Upper torso (same as active treatment)
  Interventions: Drug: Transdermal Ethinyl Estradiol/Norelgestromin Patch
- Placebo (Placebo Comparator): Placebo Transdermal Patch
  Detailed Description:
  Active Ingredients: None (placebo patch with identical appearance)
  Administration Schedule:
  1 patch applied every 7 days Total treatment duration: 21 days (3 patches total) Application Site: Upper torso (same as active treatment)
  Interventions: Drug: Placebo Patch

INTERVENTIONS:
Drug: Transdermal Ethinyl Estradiol/Norelgestromin Patch — Transdermal contraceptive patch containing ethinyl estradiol 600 micrograms and norelgestromin 6 milligrams per patch, manufactured by GEDEON RICHTER PLC and imported by Abbott.
  Other Names: Ethinyl Estradiol and Norelgestromin Transdermal Patch; Transdermal Contraceptive Patch; Combined Hormonal Contraceptive Patch; Hormonal Patch
  Arms: Treatment
Drug: Placebo Patch — Identical-appearing transdermal patches without active hormonal ingredients , manufactured and imported by Convatec.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of transdermal contraceptive patches in treating irregular vaginal bleeding in women over 18 years old who are using contraceptive implants and experiencing abnormal vaginal bleeding. The main questions it aims to answer are:

* Does transdermal ethinyl estradiol and norelgestromin patch effectively treat irregular vaginal bleeding caused by contraceptive implants compared to placebo?
* What proportion of participants will report cessation of vaginal bleeding during treatment and remain bleeding-free at day 14 of treatment?
* What is the safety profile and adherence rate of the transdermal patch treatment?

Researchers will compare participants receiving active hormonal patches (ethinyl estradiol 600 mcg + norelgestromin 6 mg) to those receiving placebo patches to see if the hormonal treatment effectively stops irregular vaginal bleeding.

Participants will:

* Apply transdermal patches for 21 days (changing patch every 7 days - total of 3 patches)
* Attend follow-up visits at days 7, 14, 21, and 3 months (day 14 in-person, others via telephone)
* Complete bleeding diaries and report any side effects
* Follow-up schedule:

Day 7: Telephone follow-up to assess bleeding pattern, side effects, and patch adherence Day 14: In-person visit at the clinic for comprehensive evaluation including bleeding assessment, side effects monitoring, and adherence check Day 21: Telephone follow-up to evaluate treatment completion, ongoing bleeding status, and need for additional treatment 3 months: Final telephone follow-up to assess long-term outcomes and recurrence of bleeding

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years and older
* Regular menstrual cycles : at least 1 cycle prior to contraceptive implant insertion
* Normal pelvic examination and transvaginal ultrasound results
* Normal cervical cancer screening within the past 3 years
* Irregular vaginal bleeding defined as: Bleeding for more than 8 consecutive days, or Bleeding-free intervals of 15 days or less

Exclusion Criteria:

* Previous treatment for irregular vaginal bleeding within the past 3 months
* Pregnancy
* Contraindications to estrogen or progestin use
* Allergy to estrogen or progestin
* Allergy to hormonal patches
* Heavy vaginal bleeding causing anemia symptoms such as: Fatigue/Fainting/Dizziness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants reporting cessation of vaginal bleeding during treatment and remaining bleeding-free at day 14 | day 14 of treatment
  The proportion of study participants who report complete cessation of abnormal vaginal bleeding while receiving the transdermal contraceptive patch treatment and continue to report no vaginal bleeding on day 14 of the 21-day treatment period.

SECONDARY OUTCOMES:
Proportion of participants with at least 7 consecutive bleeding-free days during treatment month | Throughout the treatment month (days 1-21 of treatment)
Proportion of participants reporting cessation of vaginal bleeding during treatment and remaining bleeding-free at day 7 | day 7 of treatment
Proportion of participants reporting cessation of vaginal bleeding during treatment and remaining bleeding-free at day 21 | day 21 of treatment
Number of days of treatment required before cessation of vaginal bleeding | From treatment initiation (day 1) until bleeding cessation, assessed throughout 21-day treatment period
Number of days of spotting/breakthrough bleeding during treatment | Throughout the 21-day treatment period
Number of days before recurrence of vaginal bleeding after treatment cessation | From end of treatment (day 21) until bleeding recurrence, assessed up to 3 months post-treatment
Treatment-related adverse events | Throughout treatment period (21 days) and follow-up period (3 months post-treatment)
Treatment adherence/compliance | Throughout the 21-day treatment period

CONTACTS AND LOCATIONS:
Locations (1):
- Family Planning Clinic, King Chulalongkorn Memorial Hospital, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-06): https://cdn.clinicaltrials.gov/large-docs/35/NCT07083635/Prot_SAP_000.pdf